CLINICAL TRIAL: NCT01111058
Title: Randomized Phase II Trial of Everolimus Versus Placebo as Adjuvant Therapy in Patients With Locally Advanced Squamous Cell Cancer of the Head and Neck (SCCHN)
Brief Title: Everolimus Versus Placebo in Head and Neck Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Slow accrual
Sponsor: University of Chicago (Other)
Collaborators: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 09-266-B
Record Dates: First submitted 2010-04-23; First posted 2010-04-27 (Estimated); Results first posted 2020-04-07 (Actual); Last update posted 2020-04-07 (Actual); Status verified 2020-03

CONDITIONS: Head and Neck Cancer
Keywords: Squamous Cell Cancer
MeSH Terms: conditions — Head and Neck Neoplasms; Neoplasms, Squamous Cell | interventions — Everolimus

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Everolimus (RAD001) (Experimental): Subjects will receive Everolimus 10 mg daily
  Interventions: Drug: Everolimus (RAD 001)
- Placebo (Experimental): Subjects will receive double-blind placebo
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Everolimus (RAD 001) — 10mg of Everolimus or Placebo taken by mouth once daily for 1 year or until progression (whichever comes first).
  Arms: Everolimus (RAD001)
Other: Placebo
  Arms: Placebo

SUMMARY:
Primary: Two-year progression-free (tumor does not grow or spread) survival in subjects treated with everolimus versus placebo after definitive local therapy.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Squamous cell carcinoma of the head and neck (stage IVa or IVb). No evidence (absence)of disease by scan.
* 18 years or older.
* Performance status 70% or better.
* Adequate marrow, renal and liver function (will be tested by labs). _ Able give consent.

Exclusion Criteria:

* Currently receiving anti-cancer treatment.
* Major surgery or traumatic injury within 4 weeks.
* Radiotherapy related toxicities.
* Lip, nasopharynx, nasal cavity, paranasal sinus, salivary gland, skin, or thyroid primary tumors
* Receiving other investigational drugs.
* Receiving chronic, systemic treatment with corticosteroids or another immunosuppressive agent.
* Receive immunization with attenuated live vaccines (seasonal flu shot)1 week before starting this .
* Show evidence of disease (cancer).
* Uncontrolled medical conditions such as: unstable angina, congestive heart failure, diabetes, severely impaired lung function.
* Liver disease such as cirrhosis, severe hepatic impairment, Hepatitis B or C.
* Active, uncontrolled severe infections
* Other malignancies within the past 3 years except for adequately treated carcinoma of the cervix or basal or squamous cell carcinomas of the skin.
* Known History of HIV positivity.
* Impaired gastrointestinal function that may alter absorption of Everolimus such as ulcerative disease, uncontrolled nausea, vomiting, diarrhea, malabsorption syndrome or small bowel resection.
* Patients with an active, bleeding diathesis.
* Female patients who are pregnant or breast feeding, or adults of reproductive potential who are not using effective birth control methods. )
* Male patient whose sexual partner(s) are Women of child bearing potential who are not willing to use adequate.

contraception, during the study and for 8 weeks after the end of treatment

* Patients who have received prior treatment with an mTOR inhibitor (sirolimus, temsirolimus, everolimus).
* Patients with a known hypersensitivity to Everolimus or other rapamycin analogues (sirolimus, temsirolimus) or to its excipients.
* History of noncompliance to medical regimens.
* Patients unwilling to or unable to comply with the protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2010-04; Primary Completion 2018-04 (Actual); Study Completion 2018-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tanguy Seiwert, M.D., Principal Investigator — The University of Chicago Medical Center
Locations (17):
- United States (17):
  - University of Miami, Miami, Florida
  - Northwestern University, Chicago, Illinois
  - University of Illinois-Chicago, Chicago, Illinois
  - The University of Chicago Medical Center, Chicago, Illinois
  - Ingalls Cancer Research Center, Harvey, Illinois
  - University of Kansas, Kansas City, Kansas
  - Louisianna State University, Shreveport, Louisiana
  - Tufts Medical Center, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - University of Minnesota, Minneapolis, Minnesota
  - University of Mississippi, Jackson, Mississippi
  - Washington University, St Louis, Missouri
  - University of North Carolina, Chapel Hill, North Carolina
  - Ohio State University, Columbus, Ohio
  - Medical University of South Carolina Hollings Cancer Center, Charleston, South Carolina
  - Vanderbilt University, Nashville, Tennessee
  - The University of Texas Medical Branch at Galveston, Galveston, Texas

REFERENCES:
- [Derived] Nathan CO, Hayes DN, Karrison T, Harismendy O, Flores JM, Moore-Medlin T, Vokes EE, Gutkind JS, Neupane P, Mills G, Sargi Z, Seiwert T, Grilley-Olson J, Day T, Gillison M, Wade JL, Feldman L, Jha G, Kozloff M, O'Leary M, Worden FP, Cohen EEW. A Randomized Multi-institutional Phase II Trial of Everolimus as Adjuvant Therapy in Patients with Locally Advanced Squamous Cell Cancer of the Head and Neck. Clin Cancer Res. 2022 Dec 1;28(23):5040-5048. doi: 10.1158/1078-0432.CCR-21-4290. PMID 36194164
- See also: The University of Chicago Comprehensive Cancer Center Web Page — http://uccrc.uchicago.edu/

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Subjects will receive double-blind placebo
  Placebo
Period: Overall Study
Arm/Group | Everolimus (RAD001) | Placebo
Started | 28 | 24
Completed | 28 | 24
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Everolimus (RAD001) | Placebo | Total
Number analyzed (Participants) | 28 | 24 | 52
Age, Continuous [Mean (Full Range); unit: years] | 58.0 [37 to 71] | 57.4 [37 to 76] | 57.7 [37 to 76]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 4 | 9
  Male | 23 | 20 | 43
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 3 | 6
  White | 25 | 20 | 45
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 28 | 24 | 52

OUTCOME MEASURES:

1. Primary Outcome: 2 Year Progression Free Survival Rate
Description: Time to disease progression or death from any cause--2 year rate
Time Frame: 2 years
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Everolimus (RAD001) | Placebo
Number analyzed (Participants) | 28 | 24
percentage of patients | 56.1 [31.1 to 81.2] | 55.9 [34.1 to 77.8]
Statistical Analysis 1: Comparison: Everolimus (RAD001) vs Placebo; Test type: Superiority; p = 0.90, Comparison of Kaplan-Meier estimates; Used Greenwood standard errors; Difference in survival proportions = 0.0022, 95% CI 2-sided [-0.33 to 0.33]
Statistical Analysis 2: Comparison: Everolimus (RAD001) vs Placebo; Test type: Superiority; p = 0.54, Log Rank

2. Secondary Outcome: Number of Participants With Toxicity
Description: Adverse event rate, any type, any grade regardless of attribution
Time Frame: 4 years
Measure: Count of Participants; unit: Participants
Arm/Group | Everolimus (RAD001) | Placebo
Number analyzed (Participants) | 28 | 24
Participants | 25 | 16
Statistical Analysis 1: Comparison: Everolimus (RAD001) vs Placebo; Test type: Superiority; p = 0.086, Fisher Exact

3. Secondary Outcome: Site of Progression: Local-regional
Description: Number of patients with local-regional progression
Time Frame: 4 years
Measure: Count of Participants; unit: Participants
Arm/Group | Everolimus (RAD001) | Placebo
Number analyzed (Participants) | 28 | 24
Participants | 2 | 5

4. Secondary Outcome: Site of Progression: Distant
Description: Number of patients with distant progression
Time Frame: 4 years
Measure: Count of Participants; unit: Participants
Arm/Group | Everolimus (RAD001) | Placebo
Number analyzed (Participants) | 28 | 24
Participants | 2 | 2

5. Secondary Outcome: Site of Progression: Unknown
Description: Number of patients with unknown site of progression
Time Frame: 4 years
Measure: Count of Participants; unit: Participants
Arm/Group | Everolimus (RAD001) | Placebo
Number analyzed (Participants) | 28 | 24
Participants | 1 | 1

6. Secondary Outcome: Second Primary Tumor
Description: Number of patients with second primary tumor
Time Frame: 4 years
Population: Data not systematically recorded.
Arm/Group | Everolimus (RAD001) | Placebo
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Akt/mTOR Pathway Activation
Description: mTOR positive in tumor tissue
Time Frame: Baseline
Population: Data were not collected.
Arm/Group | Everolimus (RAD001) | Placebo
Number analyzed (Participants) | 0 | 0

8. Secondary Outcome: Correlation of Akt/mTOR Status With Progression-free Survival
Description: mTOR positive in tumor tissue
Time Frame: 4 years
Population: Data were not collected.
Arm/Group | Everolimus (RAD001) | Placebo
Number analyzed (Participants) | 0 | 0

9. Secondary Outcome: Determine if PTEN Status is a Predictive Biomarker
Description: Differential effect of PTEN status on progression-free survival between the two arms
Time Frame: 4 years
Population: Data were not collected.
Arm/Group | Everolimus (RAD001) | Placebo
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 4 years
Arm/Group | Everolimus (RAD001) | Placebo
All-Cause Mortality (participants affected / at risk) | 4/28 | 4/24
Serious Adverse Events (participants affected / at risk) | 3/28 | 5/24
Other Adverse Events (participants affected / at risk) | 25/28 | 14/24
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Everolimus (RAD001) (N=28) | Placebo (N=24)
Pharyngitis (Infections and infestations) | 1 | 0
Skin infection (Infections and infestations) | 1 | 0
Thromboembolic event (Vascular disorders) | 1 | 0
Dysphagia (General disorders) | 0 | 1
Hypertension (Vascular disorders) | 0 | 1
Leukemia secondary to oncology chemotherapy (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, specify (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Suicidal ideation (Psychiatric disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Everolimus (RAD001) (N=28) | Placebo (N=24)
Abdominal pain (Gastrointestinal disorders) | 3 | 0
Alanine aminotransferase increased (Investigations) | 3 | 1
Anemia (Blood and lymphatic system disorders) | 6 | 1
Anorexia (Metabolism and nutrition disorders) | 8 | 3
Aspartate aminotransferase increased (Investigations) | 3 | 2
Cholesterol high (Investigations) | 9 | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 4 | 0
Creatinine increased (Investigations) | 2 | 1
Diarrhea (Gastrointestinal disorders) | 3 | 2
Dry mouth (Gastrointestinal disorders) | 8 | 6
Dysgeusia (Nervous system disorders) | 3 | 1
Dysphagia (Gastrointestinal disorders) | 2 | 2
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Ear pain (Ear and labyrinth disorders) | 2 | 0
Facial pain (General disorders) | 3 | 1
Fatigue (General disorders) | 7 | 4
Fever (General disorders) | 2 | 0
Headache (Nervous system disorders) | 4 | 2
Hyperglycemia (Metabolism and nutrition disorders) | 4 | 1
Hypertriglyceridemia (Metabolism and nutrition disorders) | 7 | 2
Hyponatremia (Metabolism and nutrition disorders) | 3 | 6
Infections and infestations - Other, specify (Infections and infestations) | 2 | 0
Insomnia (Psychiatric disorders) | 2 | 0
Investigations - Other, specify (Investigations) | 2 | 0
Lymphocyte count decreased (Investigations) | 9 | 1
Nausea (Gastrointestinal disorders) | 4 | 3
Neutrophil count decreased (Investigations) | 4 | 1
Pain (General disorders) | 3 | 0
Papulopustular rash (Infections and infestations) | 3 | 0
Platelet count decreased (Investigations) | 7 | 1
Rash acneiform (Skin and subcutaneous tissue disorders) | 2 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 3 | 0
Sinusitis (Infections and infestations) | 2 | 0
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 2 | 2
Skin infection (Infections and infestations) | 3 | 0
Pharyngitis (Infections and infestations) | 13 | 2
Tinnitus (Ear and labyrinth disorders) | 2 | 0
White blood cell decreased (Investigations) | 10 | 2
Hypercalcemia (Metabolism and nutrition disorders) | 0 | 2
Hypoglycemia (Metabolism and nutrition disorders) | 1 | 2
Hypophosphatemia (Metabolism and nutrition disorders) | 1 | 2
Upper respiratory infection (Investigations) | 0 | 2
Vomiting (General disorders) | 1 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2012-02-14): https://cdn.clinicaltrials.gov/large-docs/58/NCT01111058/Prot_SAP_000.pdf